CLINICAL TRIAL: NCT07202572
Title: Comparative Effects Of Virtual Reality Vs Sham VR On Fibromyalgia Impact: A Randomized Crossover Clinical Trial
Brief Title: A Study Of Virtual Reality Vs Sham VR On Fibromyalgia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anushka Irani, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 25-006773
Record Dates: First submitted 2025-09-30; First posted 2025-10-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
Keywords: Virtual Reality
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled, two-period crossover clinical trial designed to evaluate the effects of TRIPP VR meditation in individuals with fibromyalgia. Twenty participants will be randomly assigned in a 1:1 ratio to one of two intervention sequences: Sequence A will receive TRIPP VR meditation for 2 weeks, followed by a 2-week washout period, then 2 weeks of sham VR; Sequence B will receive sham VR for 2 weeks, followed by a 2-week washout period, then 2 weeks of TRIPP VR meditation. The crossover design allows each participant to serve as their own control, and the washout period is intended to minimize potential carryover effects between intervention phases.
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention type. They will not be informed whether they are receiving the active intervention (TRIPP VR meditation) or the sham VR. Study staff administering the interventions will not be blinded due to the nature of the VR content and setup requirements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sequence A (TRIPP VR to Sham VR) (Experimental): Participants in this arm will receive 2 weeks of TRIPP VR meditation followed by a 2-week washout period, then 2 weeks of sham VR.
  Interventions: Device: TRIPP VR Meditation
- Sequence B (Sham VR to TRIPP VR) (Sham Comparator): Participants in this arm will receive 2 weeks of sham VR followed by a 2-week washout period, then 2 weeks of TRIPP VR meditation.
  Interventions: Behavioral: Sham VR

INTERVENTIONS:
Device: TRIPP VR Meditation — Participants engage with the TRIPP virtual reality meditation program for 2 weeks. The TRIPP platform delivers guided mindfulness and breathing exercises through an immersive VR environment designed to promote relaxation and emotional regulation. Sessions are delivered via VR headset and used on a regular schedule (e.g., daily or as prescribed).
  Arms: Sequence A (TRIPP VR to Sham VR)
Behavioral: Sham VR — Participants engage with a sham virtual reality experience for 2 weeks. The sham VR consists of non-therapeutic, visually engaging content without meditative, guided mindfulness, or relaxation components. It is designed to mimic the immersive nature of the TRIPP VR platform without delivering active therapeutic content.
  Arms: Sequence B (Sham VR to TRIPP VR)

SUMMARY:
The purpose of this study is to understand the therapeutic impact of VR on Fibromyalgia symptoms and potentially increase the scope of treatment options for patients suffering from Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 years old
* Diagnosis of fibromyalgia based on ACR 2016 criteria
* Stable on current medications and non-pharmacologic treatments for 4 weeks
* Ability and willingness to use a Meta Quest 3 VR headset Fluent in English
* Provide informed consent

Exclusion Criteria:

* History of seizures or conditions contraindicating VR use
* Severe psychiatric illness (e.g., psychosis)
* Cognitive impairment interfering with study participation
* Participation in other interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire Revised (FIQR) Score After Sham vs. Active VR | Baseline, Week 2, and Week 4
  The primary outcome is the change in Fibromyalgia Impact Questionnaire Revised (FIQR) score from baseline to post-intervention, comparing scores after sham VR and after active TRIPP VR meditation. FIQR ranges from 0-100 and higher scores indicate higher impact of the condition, ie are worse. FIQR will be measured at baseline, week 2, and week 4. For Sequence A, the sham VR score is taken at week 4; for Sequence B, at week 2. For Sequence A, the active VR score is at week 2; for Sequence B, at week 4. The primary comparison will be the within-subject difference in FIQR change from baseline between sham and active VR periods.

CONTACTS AND LOCATIONS:
Overall Officials: Anushka Irani, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials